CLINICAL TRIAL: NCT07270380
Title: A Multi-center, Single-arm, Historically Controlled Pivotal Trial, to Assess the Safety and Effectiveness of Genex G as Part of the Surgical Treatment of Osteomyelitis of the Extremities.
Brief Title: Antibiotic Device for Osteomyelitis of the Extremities Pivotal Trial - Genex With Gentamicin.
Acronym: ADOPT GG
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Biocomposites Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201924
Record Dates: First submitted 2025-11-26; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Osteomyelitis
Keywords: Single Arm; Historical Control; Pivotal Device Study; Bone Void Filler; Gentamicin; Systemic Antibiotics; genex
MeSH Terms: conditions — Osteomyelitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Single Arm (Experimental): Participants will receive genex with Gentamicin, an antibiotic loaded bone void filler that supports bone healing, as part of the surgical treatment of osteomyelitis of the extremities.
  Interventions: Device: genex with gentamicin (genex G)

INTERVENTIONS:
Device: genex with gentamicin (genex G) — genex with gentamicin will be implanted during debridement surgery

SUMMARY:
The purpose of this trial is to determine if genex with gentamicin (genex G) an antibiotic loaded bone void filler, works to treat and is a safe option as part of the surgical treatment of osteomyelitis in the extremities.

DETAILED DESCRIPTION:
This trial is a multi-center, single arm, historically controlled, pivotal device study.

All participants diagnosed with osteomyelitis of the extremities (Cierny-Mader Classification grades I-IV) can be considered. All participants will undergo surgical debridement and will receive genex with gentamicin (genex G) antibiotic loaded bone void filler as part of the surgical treatment of osteomyelitis of the extremities. Participants will receive antibiotics per site specific requirements as clinically indicated. All participants will be followed up for 24 Months.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with osteomyelitis of the extremities (for a minimum of 6 months) that requires surgical intervention (Cierny-Mader classification of osteomyelitis grades I-IV)
2. Patients at least 18 years of age *1
3. Patient willing and able to provide written informed consent
4. Patient geographically stable and able to comply with the required follow-up visits and testing schedule as assessed by the investigator
5. Ability to achieve adequate surgical soft tissue coverage of the wound (primary tissue closure or surgical reconstruction including local and free soft tissue transfer)

   * 1 Patients between 18 and 22 years of age require confirmation of skeletal maturity as validated by radiographs of the bone to be treated.

Exclusion Criteria:

1. Renal failure or documented chronic kidney disease with serum creatinine ≥3.5 mg/dL (309umol/L) or being treated with dialysis
2. Participants with a terminal or palliative diagnosis (e.g. terminal cancer diagnosis) deemed to have less than 1 year life expectancy by their health care team
3. Uncontrolled diabetes mellitus (haemoglobin A1c levels >10%)
4. Pre-existing calcium metabolism disorder
5. Women who are pregnant or breastfeeding or planning on becoming pregnant during the study (a pregnancy test will be done in women of childbearing potential at screening and on the day of surgery)
6. History of hypersensitivity or contraindication to the investigational device or any of its ingredients (calcium phosphate, β-tricalcium phosphate, and aminoglycoside antibiotics)
7. Participation in an investigational drug/device study (within the last 60 days) or prior enrolment to the ADOPT GG study
8. Clinically significant or unstable medical or surgical condition that in the investigators opinion may preclude safe and complete study participation (for example patients medically unfit for surgery, general anaesthesia, or any risk of significant blood loss resulting in significant risk to loss of life)
9. Current untreated malignant neoplasm(s), or current treatment with radiation therapy or chemotherapy
10. Current or recent history (within last 2 years) of active substance abuse (e.g. recreational drugs, narcotics, or alcohol) that meets DSM-5 severe criteria
11. Current user of any products containing nicotine
12. Currently incarcerated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
No further requirement for antibiotic treatment due to persisting symptoms of infection at the index site (i.e., additional antibiotics prescribed following completion of the initial systemic antibiotics prescribed post surgery. | Month 12
  Further requirement for antibiotic treatment due to persisting symptoms of infection at the site of treatment will be assessed at Month 12.
No further surgical interventions required due to infection at the index site. | Month 12
  Need for further surgical interventions required due to infection at the index site will be assessed at Month 12.
No recurrence of sinus formation at the index site. | Month 12
  Recurrence of sinus formation at the index site will be assessed by a non-contrast CT scan at week 2 & Month 12. Clinical endpoint assessments will also be used to measure this at post operative follow-up visits and will be assessed at Month 12.

SECONDARY OUTCOMES:
No additional requirement for antibiotic treatment due to persisting symptoms of infection at the treatment site, i.e., additional antibiotics prescribed following completion of the initial systemic antibiotics prescribed post-surgery. | Month 24
  Further requirement for antibiotic treatment due to persisting symptoms of infection at the site of treatment will be assessed at Month 24.
No radiographic evidence of post op fractures. | Month 24
  Radiographic evidence of post-operative fractures will be evidenced by X-ray & CT evaluations and assessed at Month 24.
Radiographic evidence of new bone healing. | Month 24
  Radiographic evidence of new bone healing will be evidenced by X-ray and CT evaluations and assessed at Month 24.
No recurrence of sinus formation at the treatment site. | Month 24
  Recurrence of sinus formation at the index site will be assessed by contrast enhanced CT evaluation and Clinical endpoint assessments measured at Month 24.
No secondary surgical interventions (SSI's) related to the investigational treatment. | Month 24
  Secondary Surgical interventions (SSI's) related to the investigational treatment will be assessed at Month 24.
No serious adverse events that are definitely related to genex G. | Month 24
  Serious adverse events that are definitely related to genex G will be assessed at Month 24.
Radiographic Evidence of new bone formation and product reabsorption. | Month 24
  Radiographic evidence of new bone formation and product reabsorption will be evidenced by X-ray and CT evaluations during the course of the trial and recorded on the participants electronic case report form (eCRF).
Infection resolution evaluated by radiographic assessment and clinical endpoints. | Month 24
  Radiographic evidence of infection resolution will be evidenced by contrast enhanced CT evaluations and clinical endpoint assessments assessed during the course of the trial and recorded on the participants electronic case report form (eCRF).
Adverse events including wound problems, reaction to combination product, fracture at treatment site. | Month 24
  Adverse events including wound problems, reaction to combination product, fracture at treatment site will be assessed during the course of the trial and recorded on the participants electronic case report form (eCRF).
Secondary Surgical Interventions (SSI's) | Month 24
  Number of Secondary Surgical Interventions (SSI's) will be assessed during the course of the trial and recorded on the participants electronic case report form (eCRF).
Number of participants discontinuing therapy prematurely due to a device related event. | Month 24
  Number of participants discontinuing therapy prematurely due to a device related event will be assessed during the course of the trial and recorded on the participants electronic case report form (eCRF).
Number of hospitalisations/re-hospitalisation due to treatment site Osteomyelitis. | Month 24
  Number of hospitalisations/re-hospitalisation due to treatment site Osteomyelitis.
Quality of Life EQ-5D-5L | Month 24
  Impact on the participants Quality of Life will be measured by the EQ-5D-5L during the course of the trial and recorded on the participants electronic case report form (eCRF).

CONTACTS AND LOCATIONS:
Overall Officials: Keira Watts, PHD, Study Director — Biocomposites Ltd

IPD SHARING:
Plan to Share IPD: No